CLINICAL TRIAL: NCT01913379
Title: A Phase I Randomized, Open-label, 3-arm Parallel-design Study to Determine the Effect of Multiple-dose Gemfibrozil or Itraconazole on the Pharmacokinetics, Safety and Tolerability of Single-dose MDV3100 (ASP9785) in Healthy Male Subjects
Brief Title: Drug-drug Interaction Study With MDV3100 (ASP9785) and Gemfibrozil and Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 9785-CL-0006; 2011-000333-37 (EudraCT Number)
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Subjects; Pharmacokinetics; Drug-Drug Interaction
Keywords: Phase 1; MDV3100; Gemfibrozil; Itraconazole; Xtandi; enzalutamide
MeSH Terms: interventions — enzalutamide; Gemfibrozil; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: MDV3100 (Experimental)
  Interventions: Drug: MDV3100
- 2: MDV3100 and gemfibrozil (Experimental)
  Interventions: Drug: MDV3100; Drug: Gemfibrozil
- 3: MDV3100 and itraconazole (Experimental)
  Interventions: Drug: MDV3100; Drug: Itraconazole

INTERVENTIONS:
Drug: MDV3100 — Oral
  Other Names: ASP9785; Xtandi; enzalutamide
Drug: Gemfibrozil — Oral
  Arms: 2: MDV3100 and gemfibrozil
Drug: Itraconazole — Oral
  Arms: 3: MDV3100 and itraconazole

SUMMARY:
A study to assess possible drug-drug interactions between MDV3100 and gemfibrozil and MDV3100 and Itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of at least 65.0 kg and no greater than 85.0 kg.
* Body Mass Index (BMI) of at least 18.5 and no greater than 30.0 kg/m2.

Exclusion Criteria:

* Known or suspected hypersensitivity to MDV3100, itraconazole, gemfibrozil, any components of the formulations used, or any history of liver toxicity with other drugs.
* Confirmed CYP2C8 PM status based on genotyping analysis.
* Any of the liver function tests above the upper limit of normal. A retest to confirm the result may be performed once.
* History of seizure, including any febrile seizure, loss of consciousness, or transient ischemia attack within 12 months prior to enrollment (Day 1 visit), or any condition that may pre-dispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization).
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug (excluding non-active hay fever).
* Abnormal pulse and/or blood pressure (BP) measurements at the pre-study visit as follows: Pulse <40 or >90 bpm; mean systolic BP >140 mmHg ; mean diastolic BP >90 mmHg (BP measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically).
* A QTc interval of >430 ms after repeated measurements (consistently after duplicate measurements), a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS).
* Regular use of any inducer of metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit.
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetic profile of MDV3100 by Cmax (Maximum concentration) | Day 1 through Day 53 (29 times)
Assessment of pharmacokinetic profile of MDV3100 by AUCinf (AUC extrapolated to infinity) | Day 1 through Day 53 (29 times)
Assessment of pharmacokinetic profile of MDV3100 by AUC0-432h (AUC from the time of dosing to 432 hours post-dose) | Day 1 through Day 53 (29 times)

SECONDARY OUTCOMES:
Assessment of pharmacokinetic profile of MDV3100 | Day 1 through Day 53 (29 times)
  tmax (Time to attain Cmax), t1/2 (Apparent terminal elimination half life), Vz/F (Apparent volume of distribution during the terminal phase after extra vascular dosing) and CL/F(Apparent total body clearance after extra vascular dosing)
Assessment of pharmacokinetic profile of the metabolites MDPC0001 and MDPC0002 | Day 1 through Day 53 (29 times)
  Cmax, AUC0-432h, tmax, t1/2, and AUC0-inf
Assessment of metabolite-to-parent ratios for MDV3100 | Day 1 through Day 53 (29 times)
  This may additionally be reported to assess effects on particular enzyme pathways
Assessment of Gemfibrozil and gemfibrozil 1-O-β-glucuronide (Arm 2) | Day 1 through Day 53 (50 times)
  Cmax, C0h, Cmin, tmax, AUCtau
Assessment of itraconazole and hydroxyitraconazole (Arm 3) | Day 1 through Day 53 (50 times)
  Cmax, C0h, Cmin, tmax, AUCtau
Safety as assessed by recording adverse events, laboratory assessments, vital signs and electrocardiograms (ECGs) | Day 1 through Day 53
  In arm 3, liver function tests (AST, ALT, GGT, total bilirubin) will be done regularly during itraconazole dosing

CONTACTS AND LOCATIONS:
Overall Officials: Operation Senior Research Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- SGS, Paris, France

REFERENCES:
- [Derived] Gibbons JA, de Vries M, Krauwinkel W, Ohtsu Y, Noukens J, van der Walt JS, Mol R, Mordenti J, Ouatas T. Pharmacokinetic Drug Interaction Studies with Enzalutamide. Clin Pharmacokinet. 2015 Oct;54(10):1057-69. doi: 10.1007/s40262-015-0283-1. PMID 25929560